CLINICAL TRIAL: NCT04996875
Title: A Phase 2 Open-Label, Multicenter Clinical Study of the Safety, Efficacy, Pharmacokinetic, and Pharmacodynamic Profiles of CGT9486 as a Single Agent in Patients With Advanced Systemic Mastocytosis
Brief Title: (Apex) Bezuclastinib in Patients With Advanced Systemic Mastocytosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cogent Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGT9486-20-201; 2024-511407-42-00 (EU CTIS Number); 2021-001010-10 (EudraCT Number)
Record Dates: First submitted 2021-07-22; First posted 2021-08-09 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Advanced Systemic Mastocytosis (AdvSM); SM With an Associated Hematologic Neoplasm (SM-AHN); Mast Cell Leukemia (MCL); Aggressive Systemic Mastocytosis (ASM)
Keywords: Mastocytosis; Systemic Mastocytosis; Advanced Mastocytosis; Aggressive Mastocytosis; Hematologic Neoplasms; Mast Cell; Mast Cell Leukemia; Soft Tissue Neoplasms; Neoplasms by site; Skin Diseases; Immune Complex Diseases; Immune System Diseases; Hypersensitivity; Hematologic Diseases; Leukemia; Myeloid Leukemia; Acute Myeloid Leukemia; SM with Associated Hematologic Neoplasm; AdvSM; ASM; SM-AHN; MCL; Neoplasm; D816V; KIT D816V; AML; bezuclastinib; CGT9486; CGT; PLX; Connective Tissue Neoplasms; Urticaria Pigmentosa; High-risk myelodysplastic syndrome; Chronic myelomonocytic leukemia; Myeloproliferative neoplasm; High-risk myeloid neoplasm; High-risk MDS; MPN; High-risk MPN; Accelerated phase MPN; CMML
MeSH Terms: conditions — Mastocytosis, Systemic; Leukemia, Mast-Cell; Mastocytosis; Hematologic Neoplasms; Soft Tissue Neoplasms; Neoplasms by Site; Skin Diseases; Immune Complex Diseases; Immune System Diseases; Hypersensitivity; Hematologic Diseases; Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute; Neoplasms; Neoplasms, Connective Tissue; Urticaria Pigmentosa; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders

STUDY DESIGN:
Intervention Model Description: There are two parts to this study, including Part I, Dose Optimization, and Part II Expansion. Part II is separated into two stages.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- bezuclastinib (Experimental)
  Interventions: Drug: bezuclastinib

INTERVENTIONS:
Drug: bezuclastinib — Bezuclastinib is administered as tablets to be taken orally, continuously in 28-day cycles.
  Other Names: CGT9486; PLX9486

SUMMARY:
This is an open-label, two-part Phase 2 study investigating CGT9486 for the treatment of patients with Advanced Systemic Mastocytosis (AdvSM), including patients with Aggressive SM (ASM), SM with Associated Hematologic Neoplasm (SM-AHN), and Mast Cell Leukemia (MCL).

ELIGIBILITY:
Key Inclusion Criteria for Main Study:

1. Diagnosed with one of the following advanced mastocytosis diagnoses by Eligibility Committee

   1. Aggressive Systemic Mastocytosis (ASM)
   2. Systemic Mastocytosis with an Associated Hematologic Neoplasm (SM-AHN)
   3. Mast Cell Leukemia (MCL)
2. Measurable disease according to modified IWG-MRT-ECNM criteria. (A subset of patients inevaluble per mIWG-MRT-ECNM will be included in the study).
3. ECOG (0 to 3)
4. Have clinically acceptable local laboratory screening results (clinical chemistry, hematology) within certain limits

Key Exclusion Criteria for Main Study:

1. Persistent toxicity from previous therapy for AdvSM that has not resolved to ≤ Grade 1
2. Associated hematologic neoplasm requiring immediate antineoplastic therapy
3. Clinically significant cardiac disease
4. Known positivity for the FIP1L1 PDGFRA fusion. Patients with eosinophilia without detectable KIT D816V mutation must demonstrate lack of PDGFRA fusion mutation prior to enrollment
5. Seropositive for human immunodeficiency virus (HIV) 1 or 2, or positive for hepatitis B surface antigen or hepatitis C virus (HCV) antibody
6. History of clinically significant bleeding event within 30 days before the first dose of study drug or need for therapeutic anticoagulation on study
7. Diagnosed with or treated for malignancy other than the disease under study within the prior 3 years before enrollment
8. Received any cytoreductive therapy or any investigational agent less than 14 days, and for cladribine, interferon alpha, pegylated interferon, and any antibody therapy less than 28 days, before screening bone marrow biopsy
9. Received hematopoietic growth factor support within 14 days before the first dose of study drug
10. Received strong CYP3A4 inhibitors or inducers within 14 days or 5 drug half-lives, whichever is longer, before the first dose of study drug
11. Need for treatment with high dose steroids

Key Inclusion Criteria for Substudy Population:

Rollover Cohort

1. Demonstrate AHN progression requiring immediate AHN-directed therapy while receiving bezuclastinib
2. Demonstrated clinical benefit from bezuclastinib therapy
3. Have clinically acceptable local laboratory screening results (clinical chemistry, hematology) within certain limits

High-Risk Cohort

1. Receiving or indicated for AHN-directed therapy.
2. Diagnosed with one of the following pathologic diagnoses of SM-AHN:

   1. Myelodysplastic syndrome (MDS) that is high- or very high-risk
   2. Accelerated phase myeloproliferative neoplasm (MPN)
   3. MDS with excessive blasts in bone marrow or peripheral blood
   4. Chronic myelomonocytic leukemia-2 (CMML-2)
3. Have clinically acceptable local laboratory screening results (clinical chemistry, hematology) within certain limits.

Key Exclusion Criteria for Substudy Population:

1. Diagnosis of Philadelphia chromosome-positive malignancy
2. Diagnosis of acute myeloid leukemia (AML)
3. Appropriate for allogenic hematopoietic stem cell transplantation
4. Any contraindication to selected concomitant therapy
5. Rollover Cohort: Have not demonstrated acceptable tolerability of previous bezuclastinib therapy
6. High-Risk Cohort: Previously treated with investigational therapy for AdvSM
7. High-Risk Cohort: Previously treated with cytoreductive therapy and discontinued due to treatment-related toxicity
8. High-Risk Cohort: Received any cytoreductive therapy or any investigational agent less than 14 days, and for cladribine, interferon alpha, pegylated interferon, and any antibody therapy less than 28 days, before screening or archival bone marrow biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Part I: Identify clinically active and tolerable exposures of bezuclastinib in patients with AdvSM | 18 months
Part II: - Determine efficacy of bezuclastinib as measured by mIWG Objective Response Rate (ORR) - Confirm the exposure-response relationship of bezuclastinib | 18 months

SECONDARY OUTCOMES:
Pure Pathologic Response (PPR) | 18 months
  Months
Safety of CGT9486 as assessed by incidence of Adverse Events (AEs) | 18 months
  Incidence of AEs according to CTCAE version 5.0 or higher
To determine the effects of bezuclastinib on mutation allele burden. | 18 months
  Percentage change in KIT D816V
To determine the effects of bezuclastinib on serum tryptase. | 18 months
  Percentage change in Serum Tryptase
To assess the pharmacokinetics of bezuclastinib in subjects with AdvSM. | 18 months
  Percentage change in plasma concentrations of bezuclastinib
Change from baseline in histopathologic findings in blood and bone marrow | 18 months
  Percentage change in mast cell infiltration in the bone marrow and percentage change in eosinophilia and monocytosis in the blood
Change in spleen and liver volume by imaging | 18 months
  Percentage change
Duration of Response (DOR) | 18 months
  Months
Time to Response (TTR) | 18 months
  Months
Progression Free Survival (PFS) | 18 Months
  Months
Overall Survival (OS) | 18 months
  Months

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Easton, MD, Ph.D., Study Director — Cogent Biosciences, Inc.
Locations (42):
- United States (14):
  - University of Alabama at Birmingham (UAB) Hospital, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford Cancer Institute, Stanford, California
  - Galiz Research, Hialeah, Florida
  - Winship Cancer Institute - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - MUSC Health University Medical Center, Charleston, South Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute - University of Utah Health, Salt Lake City, Utah
- Australia (3):
  - Nepean Hospital, Kingswood, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
  - Peter MacCallum Cancer Centre, Melbourne N., Victoria
- AKH Wien, Universitatsklinikum, Vienna, Austria
- CHU de Liege, Liège, Belgium
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Michael's Hospital - Unity Health Toronto, Toronto, Ontario
- France (3):
  - Necker-Enfants Malades Hospital, Paris
  - Centre Hospitalier Universitaire (CHU) de Poitiers, Poitiers
  - Centre Hospitalier Universitaire (CHU) de Toulouse, Toulouse
- Germany (4):
  - University Hospital Aachen, Aachen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - UKSH Campus Lubeck, Lübeck
  - Universitätsklinikum Mannheim, Mannheim
- Italy (4):
  - IRCCS Azienda Ospedaliero Universitaria di Bologna, Bologna
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - AOU San Giovanni di Dio e Ruggi dAragonia, Salerno
  - Azienda Ospidaleira Universitaria Integrata Verona, Verona
- University Medical Center Groningen, Groningen, Netherlands
- Oslo University Hospital, Oslo, Norway
- Public University Hospital No. 1 in Lublin, Lublin, Poland
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
- Universitätsspital Basel, Basel, Switzerland
- United Kingdom (3):
  - Guy's Hospital - NHS Foundation Trust, London, London
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University College London Hospital - NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No